CLINICAL TRIAL: NCT03567694
Title: Randomized Double-Blind Placebo-controlled Ascending Dose FIH Study to Evaluate Single and Multiple Doses of HA115 in Healthy Volunteers and to Investigate Food Effect on Pharmacokinetics After Single Oral Doses of HA115
Brief Title: Single and Multiple Doses of HA115 and Food Effect in Healthy Adult Volunteers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision
Sponsor: Conjupro Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSPC-HA115-US-101
Record Dates: First submitted 2018-06-07; First posted 2018-06-26 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Asthma
Keywords: asthma, allergic rhinitis, HA115, CRTH2 antagonists; CT133
MeSH Terms: conditions — Asthma; Rhinitis, Allergic

STUDY DESIGN:
Intervention Model Description: The study consists of 2 parts, Part A (SAD, including fed/fasted comparison) and Part B (MAD). Part A will include an assessment of the effect of a high-fat breakfast on the absorption and PK profile of HA115, performed in 10 participants at a single dose to be selected based on SAD results and predicted to be associated with therapeutic plasma concentrations. Part B will be a randomized, double-blind, placebo controlled parallel group study of up to 3 dose levels of HA115 given once daily. The number of days of dosing will be based on the results of the PK analysis from Part A. In each cohort, 8 participants will receive active compound fasted and 2 will receive placebo in a randomized, double blind fashion. Safety observations and PK evaluations will be made. Safety data will be reviewed with the SRC prior to each dose escalation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants, principal investigator, and all other study personnel involved with participant assessments will remain blinded to the actual treatment assignments of the participants. The principal investigator will be ultimately responsible for ensuring that the integrity of the blind is maintained throughout the study and will be required to notify the sponsor in the event of any breaking of the blind for any reason. An unblinded pharmacist staff will be required at the Clinical Site to comply with the study's randomization and blinding requirements. At the Clinical Site, prior to study initiation, the principal investigator will be responsible for designating a qualified pharmacy staff to serve as the unblinded pharmacy staff in the study. Unblinded pharmacy staff may not participate in any participant assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Ascending Dose and Food effect (Experimental): This is the SAD / Food effect arm. For SAD, a total of 80 subjects will be enrolled into 8 groups of 10 subjects each; within each group, 8 will receive HA115 at a single ascending dose 10, 25, 50, 100, 200, 400, 800, 1200 mg, and 2 subjects will be placebo control. For food effect study,10 participants will be administered HA115 at a single dose to be selected based on SAD results.
  Interventions: Drug: HA115; Drug: Placebo
- Multiple Ascending Dose (Experimental): For the MAD portion, 3 dose levels will be selected based on SAD results.
  Interventions: Drug: HA115; Drug: Placebo

INTERVENTIONS:
Drug: HA115 — Test Drug
Drug: Placebo — Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled Phase 1 study of HA115 capsules administered orally to healthy adult volunteers.

DETAILED DESCRIPTION:
The study consists of 2 parts, Part A (SAD, including fed/fasted comparison) and Part B (MAD). Part A will be a randomized, double blind, placebo controlled, dose-escalating titration of up to 8 single dose levels of HA115. In each cohort, 8 participants will receive active compound and 2 will receive placebo in a randomized manner. Part A will include an assessment of the effect of a high-fat breakfast on the absorption and PK profile of HA115, performed in 10 participants at a single dose to be selected based on SAD results and predicted to be associated with therapeutic plasma concentrations.

Part B will be a randomized, double-blind, placebo controlled parallel group study of up to 3 dose levels of HA115 given once daily. The number of days of dosing will be based on the results of the PK analysis from Part A. In each cohort, 8 participants will receive active compound fasted and 2 will receive placebo in a randomized, double blind fashion. Safety observations and PK evaluations will be made. Safety data will be reviewed with the SRC prior to each dose escalation.

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy males or females, 18-55 year old, inclusive, with body mass index (BMI) between 18 and 30 kg/m2, inclusive, and body weight not less than 50 kg.
2. In good general health, free from clinically significant medical or psychiatric illness or disease (as determined by medical/surgical history, physical examination, weight, 12-lead ECG, and clinical laboratory tests).
3. with normal cardiac conduction and function at screening
4. Nonsmoker within the previous 6 months (before screening), and does not use tobacco containing, or nicotine-containing products
5. Has normal clinical chemistry, hematology, coagulation, and complete urinalysis (fasted for at least 8 hours) results at screening and Day -1
6. Has a negative urine drug screen result at screening and on Day -1.
7. For all female participants, have a negative urine pregnancy test at screening and on Day -1, and must not be breastfeeding. Female participants of childbearing potential must agree to use a protocol-approved method of non-hormonal contraception as detailed in Appendix 4 from signing of the informed consent, throughout the duration of the study and for 30 days after the last dose of study drug.
8. Male participants who are nonsterilized and sexually active with a female partner of childbearing potential must agree to use a protocol-approved method of non-hormonal contraception as detailed in Appendix 4 from signing of the informed consent, throughout the duration of the study and for 30 days after the last dose of study drug.
9. Male participants must agree to not donate sperm during the study and for 3 months (90 days) after receiving the last dose of study drug.

Key Exclusion Criteria:

1. Has a history of or current clinically significant medical illness including (but not limited to) pulmonary, cardiovascular, coagulation disorders, lipid abnormalities, gastrointestinal, immunologic, endocrine, neurologic, psychiatric, or thromboembolic disease, metabolic disturbances, or any other current physical condition that the investigator considers should exclude the participant, or that could interfere with the interpretation of the study results.
2. Has current or recent (within 6 months) history of gastrointestinal disease (except for appendectomy, inguinal/umbilical hernia), or any surgical or medical condition such as Crohn's disease or liver disease, that could potentially alter the absorption, metabolism, or excretion of the study drugs.
3. Has any clinically significant medical condition, physical examination finding, ECG abnormality, or clinically significant abnormal value for clinical chemistry, hematology, coagulation, or urinalysis at Screening or at admission to the study center, as deemed appropriate by the investigator.
4. Has any of the following (participant may rescreen once for failure to meet criteria at Screening):

   * SBP >150 mmHg at Screening stable (measured in supine position)
   * DBP of >95 mmHg at Screening stable (measured in supine position).
5. History or presence of malignancy within the past 5 years, except for adequately treated localized skin cancer (basal cell or squamous cell carcinoma), which is allowed.
6. Currently suffers from clinically significant systemic allergic disease, or has a history of significant drug allergies, including but not limited to:

   * A history of anaphylactic reaction
   * Allergic reaction due to any drug that led to significant morbidity
7. Known hypersensitivity to any component of the formulation of HA115.
8. Has donated blood or had an acute loss of blood (>500 mL) during the 3 months before study drug administration or intends to donate blood or blood products within 3 months after the completion of the study.
9. Has had an acute, clinically significant illness within 30 days prior to Day 1, or has had a recent febrile illness with an abnormal body temperature for at least 72 hours before dosing on Day 1.
10. Has a history (within the past 12 months before Screening) of drug abuse (defined as any illicit drug use), or a history of alcohol abuse (defined as alcohol consumption exceeding 14 units per week), or a positive test for drugs of abuse at Screening or upon admittance to the testing facility (Day -1) or is unwilling to abstain from alcohol and drugs of abuse throughout the study.
11. Has a smoking history during the past 6 months before Screening. This includes the use of any nicotine containing substances (e.g., nicotine patch or gum, chewing tobacco, e cigarettes), or has a positive cotinine test at Screening or Day -1, or is unwilling to abstain from these products for the duration of the study.
12. Has ever received HA115 in a previous clinical study or has used any investigational compound and/or an experimental medical device within 3 months before study drug administration.
13. If male, the participant intends to impregnate others, or donate sperm during this study or for 3 months after receiving the last dose of study drug.
14. Has inadequate venous access for the required blood draws for the study.
15. Is unable to meet or perform study requirements or has a known or suspected inability to comply with the study protocol.
16. Is unable or unwilling to eat provided food (e.g., vegetarian, kosher, lactose intolerant dietary requirements).
17. Is an immediate family member of the investigator, or an employee of the study center with direct involvement in the proposed study or other studies under the direction of the investigator or study center or is in a dependent relationship with a study site employee who is involved in the conduct of this study (eg, spouse, parent, child, sibling), or may consent under duress.
18. Has been on a significantly abnormal diet during the 4 weeks preceding the first dose of study medication.
19. Has participated in another clinical trial within 60 days prior to the first dose of study medication.
20. Use of any over-the-counter (OTC) medication (including nutritional or dietary supplements, herbal preparations, or vitamins) within 7 days prior to the first dose of study medication until the end of study visit without evaluation and approval by the investigator.
21. Use of any prescription medication from 14 days prior to the first dose of study medication until the end-of-study visit.
22. Has been treated with any known drugs that are moderate or strong inhibitors/inducers of cytochrome P450 (CYP) enzymes (e.g., barbiturates, phenothiazines, cimetidine, carbamazepine) within 30 days prior to the first dose of study medication, and that, in the investigator's judgment, may impact participant safety or the validity of the study results.
23. Engagement in strenuous exercise from 48 hours prior to the first dose of study medication until the end-of-study visit.
24. Consumption of beverages or foods that contain alcohol, grapefruit, poppy seeds, broccoli, Brussel sprouts, pomegranate, star fruit, char-grilled meat, or caffeine/xanthine from 48 hours prior to the first dose of study medication until the end of study visit. P25. Is a female participant with a positive pregnancy test result.
25. Has a positive test for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus (HIV) at screening or has been previously treated for hepatitis B, hepatitis C, or HIV infection.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-10-10 (Estimated); Study Completion 2022-10-12 (Estimated)

PRIMARY OUTCOMES:
Adverse event (AE) | 36 days
  Percentage of subjects experiencing adverse event (AE).

CONTACTS AND LOCATIONS:
Overall Officials: Study Officials, Study Director — Conjupro Biotherapeutics, Inc.
Locations (1):
- CNS Network, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: No